CLINICAL TRIAL: NCT05432362
Title: ESAN II - Energy Sensing in Depression. Effects of Aronia Melanocarpa on Immunomodulation in Patients With Obesity, Depression, and Normal Weight Controls.
Brief Title: ESAN II - Energy Sensing in Depression
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ESANII
Record Dates: First submitted 2022-06-13; First posted 2022-06-27 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Immune System Tolerance; Depression; Obesity; Microbial Colonization; Diet, Healthy
Keywords: polyphenols; Aronia melanocarpa; immunomodulation; plant based food; natural food
MeSH Terms: conditions — Depression; Obesity; Communicable Diseases

STUDY DESIGN:
Intervention Model Description: This monocentric study is a food product study (comparison between in trade available polyphenol-rich juice and a placebo).
  Aronia juice is a locally produced, commercially available natural source of various secondary plant nutrients. It naturally contains high amounts of polyphenols. The placebo juice is prepared according to a published recipe and contains comparable amounts of nutrients such as vitamins and minerals but is totally polyphenol-free.
  Six study groups are designated:
  Group VN = normal weight participants receiving polyphenol-rich juice (verum) (n=20) Group VA = adipose participants receiving polyphenol-rich juice (verum) (n=20) Group VD = depressive patients receiving polyphenol-rich juice (verum) (n=20) Group CN = normal weight participants receiving placebo (control) (n=20) Group CA = adipose participants receiving placebo (control) (n=20) Group CD = depressive patients receiving placebo (control) (n=20)
Who Masked: Participant
Masking Description: The randomizer (online tool of the Medical University of Graz) will be used for randomisation of group assignment. The two juices are provided in the same containers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Verum Normal Weight (Experimental): Normal weight participants receiving polyphenol-rich Aronia juice (verum) (n=20) The aronia juice is derived from a local producer, a common food and commercially available.
  Interventions: Other: Aronia Juice
- Verum Obesity (Experimental): Adipose participants receiving polyphenol-rich Aronia juice (verum) (n=20) The aronia juice is derived from a local producer, a common food and commercially available.
  Interventions: Other: Aronia Juice
- Verum Depression (Experimental): Depressive participants receiving polyphenol-rich Aronia juice (verum) (n=20) The aronia juice is derived from a local producer, a common food and commercially available.
  Interventions: Other: Aronia Juice
- Placebo Normal Weight (Placebo Comparator): Normal weight participants receiving placebo (control) (n=20)
  The placebo drink is prepared according to a published recipe and contains nutrients such as sugars, vitamins and minerals. It has a comparable nutrients profile as the aronia juice but is completely polyphenol-free.
  Interventions: Other: Placebo
- Placebo Obesity (Placebo Comparator): Obese participants receiving placebo (control) (n=20)
  The placebo drink is prepared according to a published recipe and contains nutrients such as sugars, vitamins and minerals. It has a comparable nutrients profile as the aronia juice but is completely polyphenol-free
  Interventions: Other: Placebo
- Placebo Depression (Placebo Comparator): Depressive participants receiving placebo (control) (n=20)
  The placebo drink is prepared according to a published recipe and contains nutrients such as sugars, vitamins and minerals. It has a comparable nutrients profile as the aronia juice but is completely polyphenol-free
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Aronia Juice — The intervention is based an the additional consumption of 200 ml natural juice a day for a period of six weeks. The participants are asked to drink the natural and commercially available juice in addition to their regular diet. Further, they are asked not to change their diets and lifestyle behaviour during the intervention.
  Arms: Verum Depression; Verum Normal Weight; Verum Obesity
Other: Placebo — A beverage is prepared according to a known recipe. It contains macro- and micronutrients in comparable amounts like the aronia juice. It is completely polyphenol free.
  Arms: Placebo Depression; Placebo Normal Weight; Placebo Obesity

SUMMARY:
The purpose of this study is to assess the effects of polyphenols from natural aronia juice on the immune system.

Therefore, the study aims to distinguish the effects of natural juices that are rich in phytonutrients such as polyphenols and carotenoids in healthy and depressive subjects in order to use the known positive effects of these food sources in the therapeutic setting.

The consumption of natural fruit juices that are rich in polyphenols and carotenoids mirror a model of vegetarian diet due to the increased micronutrient density derived from plant food. Results obtained here can be seen as preliminary explanation models for the beneficial effects of vegetarian diet.

It is hypothesized, that the consumption of naturally polyphenol rich aronia juice changes the expression of regulatory T cells, specific cells of the immune system that contribute to immunomodulation. Furthermore, beneficial changes in the gut microbiome, the metabolome and the nutritional status are expected in the studied groups.

The study was registered retrospectively (after start of recruitment) on Clinicaltrials.gov.

ELIGIBILITY:
Inclusion Criteria:

1. Socio-demographic criteria:

   1. Gender: female
   2. Age: 18-40 years
2. Confirmation of the study settings

   1. receives of information on

      * the aims,
      * methods,
      * anticipated benefits,
      * potential risks, and
      * entailed discomforts of the study
   2. signed declaration of consent
3. Subgroup of depressive patients:

   1. diagnosis of depression according to the ICD-10 criteria for depression
   2. diagnosed by an experienced psychiatrist

      * a structured diagnostic interview
      * voluntarily agreement to participate
      * signed informed consent
4. Subgroup of normal weight participants:

   * WHO criteria for normal weight (body mass index (BMI) 18.5-24.99 kg/m2)
5. Subgroup of obese participants

   * WHO criteria for obesity (BMI < 30.0 kg/m2)

Exclusion Criteria:

1. Formal criteria:

   * lack of informed consent
2. Health criteria

   1. alcohol- or drug abuse
   2. major cognitive deficits (which do not allow adequate testing)

      * according to Mini Mental Status Examination (MMSE) <20
   3. patients which are currently in the locked ward of the clinic
   4. acute or chronic diseases or infections within the previous two months

      * upper respiratory tract infections
      * fever
      * chronic inflammatory disorders
      * autoimmune-disorders
      * blood diseases
      * mitochondrial diseases
3. Digestive disorders

   1. fructose intolerance
   2. history of digestive diseases such as

      * inflammatory bowel disease
      * irritable bowel syndrome
   3. treatment that may has influenced the microbiome

      * antibiotic or antifungal treatment within the previous two months
      * daily or irregular intake of prebiotics or probiotics within the previous two months (the intake of yoghurt and dairy products are permitted)
   4. history of gastrointestinal surgery (other than appendectomy)
4. Pregnancy and period of breastfeeding

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-02-25 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Change of baseline regulatory T cells (Tregs) at 6 weeks (after the intervention) | Determination at baseline (day 0) and after 6 weeks (after the intervention)
  Tregs are involved in modulating the immune system and maintaining tolerance to self-antigens and preventing autoimmune diseases.
  Regulatory T cells (Treg) will be quantified using multiparameter flow cytometry. Monoclonal antibodies specific for surface markers such as CD3, CD4, CD45RA, CD39 and CD25 will be combined with intracellular anti-Foxp3 for the identification of human Treg.
Change of baseline regulatory T cells (Tregs) at 12 weeks (after the intervention and another 6 weeks of wash out) | Determination at baseline and after 12 weeks (after the 6-weeks intervention and another 6 weeks of wash out)
  Tregs are involved in modulating the immune system and maintaining tolerance to self-antigens and preventing autoimmune diseases. The assessment of Tregs after 12 weeks aims to identify any persisting effects of the intervention.

SECONDARY OUTCOMES:
Change of baseline gut microbiome at 6 weeks (after the intervention) | Determination at baseline (day 0) and after 6 weeks (after the intervention)
  Stool samples will be collected with the PSP spin stool DNA stool collection kit (Stratec, Birkenfeld, GER) and processed according to the suppliers recommendations. Subsequently to DNA extraction the variable V1-V2 region of the bacterial 16S rRNA gene is amplified with PCR using oligonucleotide primers BSF8 and BSR357.
Change of baseline gut microbiome at 12 weeks (after the 6-weeks intervention and another 6 weeks of wash out) | Determination at baseline and after 12 weeks (after the 6-weeks intervention and another 6 weeks of wash out)
  Stool samples will be collected with the PSP spin stool DNA stool collection kit (Stratec, Birkenfeld, GER) and processed according to the suppliers recommendations. Subsequently to DNA extraction the variable V1-V2 region of the bacterial 16S rRNA gene is amplified with PCR using oligonucleotide primers BSF8 and BSR357. The assessment of the change in the gut microbiome after 12 weeks aims to identify any persisting effects of the intervention.

OTHER OUTCOMES:
Change of baseline metabolome at 6 weeks (after the intervention) | Determination at baseline (day 0) and after 6 weeks (after the intervention)
  The metabolome can be identified in various biological materials such as blood (EDTA and serum) Metabolites in blood will be analyzed by using 1H-NMR spectra. A non-targeted approach will be applied to characterize a potential shift in the participants' metabolic profile.
Change of baseline metabolome at 12 weeks (after the 6 weeks intervention and another 6 weeks of wash out) | Determination at baseline and after 12 weeks (after the 6-weeks intervention and another 6 weeks of wash out)
  The metabolome can be identified in various biological materials such as blood (EDTA and serum) Metabolites in blood will be analyzed by using 1H-NMR spectra. A non-targeted approach will be applied to characterize a potential shift in the participants' metabolic profile.The assessment of the change in the metabolome after 12 weeks aims to identify any persisting effects of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Holasek, Prof., Principal Investigator — Medical Universtiy of Graz
Locations (1):
- Medical Universtiy of Graz, Graz, Styria, Austria

REFERENCES:
- [Background] Meyrel M, Varin L, Detaint B, Mouaffak F. [The intestinal microbiota: A new player in depression?]. Encephale. 2018 Feb;44(1):67-74. doi: 10.1016/j.encep.2017.03.005. Epub 2017 Apr 24. French. PMID 28438331
- [Background] Koopman M, El Aidy S; MIDtrauma consortium. Depressed gut? The microbiota-diet-inflammation trialogue in depression. Curr Opin Psychiatry. 2017 Sep;30(5):369-377. doi: 10.1097/YCO.0000000000000350. PMID 28654462
- [Background] De Rosa V, Galgani M, Santopaolo M, Colamatteo A, Laccetti R, Matarese G. Nutritional control of immunity: Balancing the metabolic requirements with an appropriate immune function. Semin Immunol. 2015 Sep;27(5):300-9. doi: 10.1016/j.smim.2015.10.001. Epub 2015 Oct 29. PMID 26527507
- [Background] Abella V, Scotece M, Conde J, Pino J, Gonzalez-Gay MA, Gomez-Reino JJ, Mera A, Lago F, Gomez R, Gualillo O. Leptin in the interplay of inflammation, metabolism and immune system disorders. Nat Rev Rheumatol. 2017 Feb;13(2):100-109. doi: 10.1038/nrrheum.2016.209. Epub 2017 Jan 5. PMID 28053336
- [Background] Perez-Perez A, Vilarino-Garcia T, Fernandez-Riejos P, Martin-Gonzalez J, Segura-Egea JJ, Sanchez-Margalet V. Role of leptin as a link between metabolism and the immune system. Cytokine Growth Factor Rev. 2017 Jun;35:71-84. doi: 10.1016/j.cytogfr.2017.03.001. Epub 2017 Mar 4. PMID 28285098
- [Background] Bettelli E, Carrier Y, Gao W, Korn T, Strom TB, Oukka M, Weiner HL, Kuchroo VK. Reciprocal developmental pathways for the generation of pathogenic effector TH17 and regulatory T cells. Nature. 2006 May 11;441(7090):235-8. doi: 10.1038/nature04753. Epub 2006 Apr 30. PMID 16648838
- [Background] Kim W, Lee H. Advances in nutritional research on regulatory T-cells. Nutrients. 2013 Oct 28;5(11):4305-15. doi: 10.3390/nu5114305. PMID 24169507
- [Background] Kim YS, Sayers TJ, Colburn NH, Milner JA, Young HA. Impact of dietary components on NK and Treg cell function for cancer prevention. Mol Carcinog. 2015 Sep;54(9):669-78. doi: 10.1002/mc.22301. Epub 2015 Apr 1. PMID 25845339
- [Background] Xue Z, Li D, Yu W, Zhang Q, Hou X, He Y, Kou X. Mechanisms and therapeutic prospects of polyphenols as modulators of the aryl hydrocarbon receptor. Food Funct. 2017 Apr 19;8(4):1414-1437. doi: 10.1039/c6fo01810f. PMID 28287659
- [Background] Shanahan F, van Sinderen D, O'Toole PW, Stanton C. Feeding the microbiota: transducer of nutrient signals for the host. Gut. 2017 Sep;66(9):1709-1717. doi: 10.1136/gutjnl-2017-313872. Epub 2017 Jun 29. PMID 28663354
- [Background] Vauzour D, Rodriguez-Mateos A, Corona G, Oruna-Concha MJ, Spencer JP. Polyphenols and human health: prevention of disease and mechanisms of action. Nutrients. 2010 Nov;2(11):1106-31. doi: 10.3390/nu2111106. Epub 2010 Nov 8. PMID 22254000
- [Background] Mullan A, Delles C, Ferrell W, Mullen W, Edwards CA, McColl JH, Roberts SA, Lean ME, Sattar N. Effects of a beverage rich in (poly)phenols on established and novel risk markers for vascular disease in medically uncomplicated overweight or obese subjects: A four week randomized placebo-controlled trial. Atherosclerosis. 2016 Mar;246:169-76. doi: 10.1016/j.atherosclerosis.2016.01.004. Epub 2016 Jan 6. PMID 26797134
- [Background] Aguirre L, Fernandez-Quintela A, Arias N, Portillo MP. Resveratrol: anti-obesity mechanisms of action. Molecules. 2014 Nov 14;19(11):18632-55. doi: 10.3390/molecules191118632. PMID 25405284
- [Background] Chrubasik C, Li G, Chrubasik S. The clinical effectiveness of chokeberry: a systematic review. Phytother Res. 2010 Aug;24(8):1107-14. doi: 10.1002/ptr.3226. PMID 20572194
- [Result] Morkl S, Lackner S, Muller W, Gorkiewicz G, Kashofer K, Oberascher A, Painold A, Holl A, Holzer P, Meinitzer A, Mangge H, Holasek S. Gut microbiota and body composition in anorexia nervosa inpatients in comparison to athletes, overweight, obese, and normal weight controls. Int J Eat Disord. 2017 Dec;50(12):1421-1431. doi: 10.1002/eat.22801. Epub 2017 Nov 13. PMID 29131365
- [Derived] Lackner S, Mahnert A, Moissl-Eichinger C, Madl T, Habisch H, Meier-Allard N, Kumpitsch C, Lahousen T, Kohlhammer-Dohr A, Morkl S, Strobl H, Holasek S. Interindividual differences in aronia juice tolerability linked to gut microbiome and metabolome changes-secondary analysis of a randomized placebo-controlled parallel intervention trial. Microbiome. 2024 Mar 9;12(1):49. doi: 10.1186/s40168-024-01774-4. PMID 38461313